CLINICAL TRIAL: NCT04741074
Title: A RAndomized trIal Examining the Effect of Subcutaneous Semaglutide on Kidney Transplant Candidacy for Patients With Stage 4-5 CKD or Dialysis-dependent ESKD
Brief Title: Effect of Subcutaneous Semaglutide on Kidney Transplant Candidacy
Acronym: RAISE-KT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Alexander Chang, Assistant Professor, Clinical Research, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-1050; Universal Trial Number (Registry Identifier: U1111-1249-8833)
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: CKD; Diabetic Kidney Disease; Type 2 Diabetes Mellitus in Obese; Obesity; Severe Obesity
Keywords: ckd; obesity; kidney transplant; transplant wait list; diabetic kidney disease; glp-1; semaglutide
MeSH Terms: conditions — Diabetic Nephropathies; Obesity; Obesity, Morbid; Renal Insufficiency, Chronic | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a placebo-controlled double-blind clinical trial. Study investigators and participants will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Active Comparator): This arm will receive semaglutide.
  Interventions: Drug: Semaglutide 2 mg/1.5 ml (1.34 mg/ml), prefilled pen-injector for subcutaneous injection solution
- Placebo (Placebo Comparator): This arm will receive placebo.
  Interventions: Drug: Placebo 1.5 ml, prefilled pen-injector for subcutaneous injection solution

INTERVENTIONS:
Drug: Semaglutide 2 mg/1.5 ml (1.34 mg/ml), prefilled pen-injector for subcutaneous injection solution — Dose will be started at 0.25 mg per week. Dose escalation will occur every 4 weeks to mitigate risk of gastrointestinal side effects to a maximum dose of 1.0 mg per week.
  Other Names: semaglutide
  Arms: Semaglutide
Drug: Placebo 1.5 ml, prefilled pen-injector for subcutaneous injection solution — Matched placebo solution for injection will be provided by Novo Nordisk in a 1.5 ml pre-filled pen-injector for subcutaneous injection with the same instructions on dose escalation.
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This randomized study evaluates the effect of subcutaneous semaglutide /in combination with lifestyle counseling in patients with type 2 diabetes mellitus (T2DM), overweight/obesity, and stage 4-5 chronic kidney disease (CKD) or dialysis-dependent end-stage kidney disease (ESKD) on patients' eligibility for kidney transplantation at the end of 9 months.

DETAILED DESCRIPTION:
Transplant policies regarding listing consider uncontrolled diabetes and severe obesity to be contraindications though there is great variability for exact BMI (35-45 kg/m2) and A1c (9-10%) thresholds for listing by center. Glucagon-lowering peptide-1 receptor agonists (GLP-1 RAs) offer great promise in this population as they have been shown to reduce weight, central adiposity, A1c, and risk of cardiovascular outcomes with similar effects in patients with and without CKD.

In this double-blind, placebo-controlled randomized controlled trial, the investigators will evaluate the effect of subcutaneous semaglutide 1.34 mg/ml (up to 1.0 mg per week) in combination with lifestyle counseling in patients with T2DM, overweight/obesity, and stage 4-5 CKD or dialysis-dependent ESKD on patients' eligibility for kidney transplantation in terms of diabetes control (A1c <9%) and obesity (BMI <35 kg/m2 or 35-40 kg/m2 with waist circumference <120 cm) at the end of 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. - Age ≥ 18 years
2. - BMI 25-45 kg/m2
3. - T2DM
4. - Advanced CKD* (last eGFR <30 ml/min/1.73m2 in EHR or ESKD on dialysis prior to screening) or stage G3B/A2-3 CKD (eGFR 30 to <45 ml/min/1.73m2 with albumin/creatinine ratio >30 mg/g).
5. - Fulfill kidney transplant listing criteria except for one or more of the following reasons (1: uncontrolled diabetes [A1c ≥9%); 2: severe obesity (BMI ≥ 40 kg/m2 or BMI 35-40 kg/m2 with waist circumference >120 cm). See exclusion criteria for general contraindications used for transplant listing used by majority of U.S. transplant centers].
6. - Ability to provide informed consent before any trial-related activities
7. - Access to a telephone

   * The cause of the CKD does not need to be due specifically to diabetes

Exclusion Criteria (General contraindications used for transplant listing used by majority of U.S. transplant centers)

1. - Active malignancy
2. - History of pancreatitis
3. - Active substance abuse
4. - Severe COPD
5. - Pulmonary fibrosis
6. - Symptomatic angina or recent myocardial infarction within 6 months
7. - Severe peripheral vascular disease
8. - Cirrhosis
9. - New York Health Association (NYHA) Class III-IV congestive heart failure
10. - Severe cognitive impairment
11. - Drug addiction
12. - History of non-adherence to therapy
13. - Active infection
14. - Expected life expectancy < 5 years

    Additional exclusion criteria
15. - Type 1 diabetes mellitus
16. - History of diabetic ketoacidosis within the last 12 months
17. - Planning on undergoing bariatric surgery in next 9 months.
18. - Pregnant, breast-feeding, or planned pregnancy prior to the end of participation or not using adequate contraceptive measures
19. - Self-reported average consumption of > 21 alcoholic beverages per week or binge drinking
20. - Psychiatric hospitalization in past year
21. - Principal investigator discretion (i.e. concerns about safety, compliance)
22. - Known or suspected allergy to trial medication
23. - Previous participation (i.e. randomized) in this trial
24. - Use of GLP1-RA or pramlintide within 90 days prior to screening
25. - Use of metformin (contraindicated with eGFR < 30 ml/min/1.73m2)
26. - Use of DPP-4 inhibitors within 30 days prior to screening
27. - Personal or family history of medullary thyroid cancer, multiple endocrine neoplasia types 2A and 2B syndrome
28. - Last hemoglobin A1c ≥ 12% or A1c <6% (to avoid risk of hypoglycemia) prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex R Chang, MD, MS, Principal Investigator — Geisinger Clinic
Locations (2):
- United States (2):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the time of publication of the main trial results and will be publicly available indefinitely.
Access Criteria: The deidentified IPD will be publicly available without restrictions.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Semaglutide | Placebo
Started | 7 | 8
Completed | 5 | 7
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study terminated prematurely | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Placebo | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 62.29 (3.00) | 59.13 (14.88) | 60.60 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] | 6.8 (0.38) | 6.70 (0.50) | 6.75 (0.31)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 39.7 (5.37) | 40.20 (4.12) | 39.95 (4.57)
Waist circumference [Mean (Standard Deviation); unit: cm] | 132.37 (5.99) | 124.20 (9.77) | 128.01 (13.16)

OUTCOME MEASURES:

1. Primary Outcome: Kidney Transplant Eligibility
Description: Proportion either listed for kidney transplant at 9 months or meeting the following kidney transplant candidacy criteria for A1c (<9%) and obesity (BMI <35 kg/m2 or BMI 35-40 kg/m2 with waist circumference <120 cm)
Time Frame: Ascertained at the end of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 5 | 7
Participants | 3 | 2

2. Secondary Outcome: Change in Hemoglobin A1c (HgbA1c)
Description: HgbA1c will be collected using routine procedures and measured on the same day at the central Geisinger laboratory by Turbidimetric inhibition immunoassay.
Time Frame: From baseline to 9 months
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 5 | 7
Percentage of glycosylated hemoglobin | -1.10 (1.03) | 0.33 (0.78)

3. Secondary Outcome: Change in BMI
Description: Weight will be measured at each study visit in light clothing without shoes by trained, certified staff using a calibrated, digital scale. Scales will be calibrated annually. Height will be measured at the initial study visit to the nearest 0.1 cm using a calibrated, wall-mounted stadiometer without shoes on a firm, level surface, with head in the horizontal plane.
Time Frame: From baseline to 9 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 5 | 7
kg/m^2 | -2.55 (4.25) | -.07 (2.70)

4. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference will be measured at each study visit to the nearest 0.1 cm using a Gulick II tape measure.
Time Frame: From baseline to 9 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 5 | 7
cm | -0.52 (14.38) | 3.91 (6.32)

5. Secondary Outcome: Change in Waist-to-hip Ratio
Description: Hip circumference will also be measured to the nearest 0.1 cm using a Gulick II tape measure, and waist-to-hip ratio will be calculated.
Time Frame: From baseline to 9 months
Measure: Mean (Standard Deviation); unit: cm/cm
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 5 | 7
cm/cm | -.00 (0.11) | 0.03 (0.05)

6. Secondary Outcome: Change in Body Fat Percentage
Description: Measured using bioelectrical impedance analysis
Time Frame: From baseline to 9 months
Measure: Mean (Standard Deviation); unit: Body fat percentage
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 6 | 5
Body fat percentage | -2.70 (1.93) | 0.13 (3.98)

7. Secondary Outcome: New Activation on the Transplant List
Description: Proportion of participants who were newly added to a transplant list during study period. Assessed by Geisinger kidney transplant committee (blinded to randomization assignment, independent of investigators)
Time Frame: Assessed at end of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 5 | 7
Participants | 3 | 0

8. Secondary Outcome: Receipt of Kidney Transplant
Description: Confirmed by review of electronic health record (EHR)
Time Frame: Assessed at end of 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 5 | 7
Participants | 0 | 0

9. Other Pre Specified Outcome: Change in Low-Density Lipoprotein (LDL)
Description: Collected at a Geisinger lab using routine procedures and measured on the same day at the central Geisinger laboratory by spectrophotometry.
Time Frame: Baseline to 9 months
Population: One patient in the placebo arm did not complete follow-up LDL measurement, and thus there is 1 less participant analyzed in the placebo arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 5 | 6
mg/dL | -6.20 (17.37) | -6.17 (53.63)

10. Other Pre Specified Outcome: Change in Triglycerides
Description: as for outcome 9
Time Frame: Baseline to 9 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Systolic Blood Pressure
Description: Automated office blood pressure (AOBP) will be measured (attended) using the OMRON 907-XL machine, with a 5-minute rest period in the seated position, followed by 3 measurements separated by 1-minute time intervals by trained research staff. Mid-arm circumference will be measured, and a cuff of appropriate size will be identified and the same size cuff will used for both visits.
Time Frame: Baseline to 9 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Diastolic Blood Pressure
Description: as for outcome 11
Time Frame: Baseline to 9 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Albuminuria Among Subset of Participants Without End-stage Kidney Disease
Description: Testing at the central Geisinger laboratory, using immunoturbidimetry (albumin) and Jaffe/Enzymatic (Urine Creatinine)
Time Frame: Baseline to 9 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Estimated Glomerular Filtration (eGFR) Rate Among Subset of Participants Without End-stage Kidney Disease
Description: Testing at central Geisinger lab; Creatinine-based CKD-EPI equation
Time Frame: Baseline to 9 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: All-cause Hospitalizations
Description: Collected using Geisinger EHR data
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Cardiovascular Disease (CVD) Events
Description: Collected using Geisinger EHR data using ICD codes for CVD-related hospitalizations
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Proportion Experiencing Doubling of Creatinine or End-stage Kidney Disease
Description: Collected using Geisinger EHR data using ICD codes
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Proportion Experiencing Death
Description: Collected using Geisinger EHR data
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Proportion Experiencing Gastrointestinal Disorders
Description: Assessed at each study visit
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Proportion Experiencing Gallbladder Disorders
Description: Assessed at each study visit
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Proportion Experiencing Neoplasms
Description: Assessed at each study visit
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Proportion Experiencing Hepatic Events
Description: Assessed at each study visit
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Proportion Experiencing Allergic Reactions
Description: Assessed at each study visit
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Proportion Experiencing Injection-site Reactions
Description: Assessed at each study visit
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Proportion Experiencing Hypoglycemia Events
Description: Assessed at each study visit
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Proportion Experiencing Acute Pancreatitis Events
Description: Assessed at each study visit
Time Frame: Entire 9-month study period
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 9 months
Description: Safety outcomes specifically assessed at each study visit systematically included: gastrointestinal disorders, gallbladder disorders, neoplasms, hepatic events, allergic reactions, injection-site reactions, hypoglycemia events, and acute pancreatitis events.
Arm/Group | Semaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/8
Other Adverse Events (participants affected / at risk) | 5/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=7) | Placebo (N=8)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Uremia (Renal and urinary disorders) | 1 (1) | 1 (1)
Hypertensive urgency (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=7) | Placebo (N=8)
Hypoglycemia events (Endocrine disorders) | 3 (3) | 4 (4)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (5) | 2 (2)
Gallbladder disorders (Hepatobiliary disorders) | 0 (0) | 0 (0)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0)
Hepatic events (Hepatobiliary disorders) | 0 (0) | 0 (0)
Allergic reactions (Immune system disorders) | 0 (0) | 0 (0)
Injection-site reactions (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Acute pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0)
Anemia or bleeding disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the funder due to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT04741074/Prot_SAP_000.pdf